CLINICAL TRIAL: NCT07112040
Title: Adaptation of a Intervention Protocol for Acute Post-Traumatic Stress Symptoms in Survivors of Sexual Violence: Design, Implementation, and Effectiveness in Specialized Intervention Centers
Brief Title: The Effectiveness of a Brief Early Intervention of Acute Stress Syndrome Stabilization Protocol for Victims of Sexual Violence (ASSYST-SV).
Acronym: ASSYST-SV
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Collaborators: EMDR Europe (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ASSYST-SV PROTOCOL
Record Dates: First submitted 2025-08-01; First posted 2025-08-08 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Acute Stress Symptoms; Sexual Violence
Keywords: ASSYST protocol; Acute stress; trauma; individual intervention; survivors of sexual violence
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: This is a single-arm, pre-post intervention study designed to evaluate the effectiveness of the ASSYST-VS protocol in reducing acute stress symptoms in women who have experienced sexual violence. Due to ethical considerations-given the high risk of psychopathology following sexual victimization-no control or waitlist group is included.
  Assessments are conducted at three time points: prior to the intervention (baseline), immediately after the intervention (post-treatment), and at a 3-month follow-up. The primary outcome is the reduction of acute stress symptoms. Complementary outcomes include levels of anxiety, sleep disturbances, overall mental well-being, and functional impairment.
  This design allows for an ethically sensitive, real-world evaluation of a brief, trauma-focused intervention in a vulnerable population.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ASSYST-VS Intervention (Experimental): This is a single-arm study. All participants will receive the ASSYST-SV intervention, a brief, trauma-focused psychological protocol adapted for adult women who have experienced sexual violence within the previous six months. No waitlist or control condition is included due to ethical considerations.
  Interventions: Behavioral: Behavioral - ASSYST-VS Protocol

INTERVENTIONS:
Behavioral: Behavioral - ASSYST-VS Protocol — The ASSYST-SV protocol consists of three sessions, each lasting approximately 90 minutes, ideally delivered once per week over a three-week period.
  The intervention includes:
  Session 1: Psychoeducation: Explanation of typical responses to sexual trauma, providing information about the recovery process, and establishing a strong therapeutic alliance between the client and therapist.
  Sessions 1-3: Emotional self-regulation using trauma-sensitive yoga exercises adapted for survivors of sexual violence.
  Sessions 2-3: Trauma desensitization using EMDR-informed techniques, including bilateral stimulation and self-applied tools such as the Butterfly Hug.
  Safety procedures and closure are included in all sessions to ensure emotional containment and promote participant well-being.
  The intervention is delivered by trained professionals in specialized support services for victims of gender-based violence.

SUMMARY:
TThe main objectives of this research project are twofold: (1) to conduct a narrative review of the scientific literature on the efficacy and effectiveness of psychological interventions for reducing acute post-traumatic stress symptoms in survivors of sexual violence, and to provide a solid theoretical framework on the consequences of sexual victimization and the use of EMDR interventions in this population; and (2) to develop and test an adapted version of the ASSYST protocol of Jarero´s team for survivors of sexual violence (ASSYST-SV), evaluating its effectiveness and feasibility in reducing acute stress symptoms in women who have experienced sexual violence.

This is an exploratory quasi-experimental study with a single-group pre-post design and follow-up assessments. The intervention will be delivered to women receiving care in specialized services for survivors of gender-based violence in Catalonia and Madrid. Assessments will be conducted at three time points: pre-intervention, post-intervention, and three-month follow-up. Data will be collected through a combination of clinician-administered and self-report questionnaires.

This trial is part of a larger research project (NCT05619822) that includes several related studies. Each study addresses a specific population and/or intervention, but all share the overarching aim of examining the efficacy of a comprehensive third-generation protocol for individuals with comorbid trauma and other mental health conditions.

DETAILED DESCRIPTION:
Sexual violence is associated with a high risk of developing post-traumatic stress disorder (PTSD), emotional distress, sleep disturbances, and impairments in daily functioning. Despite these risks, few interventions are tailored to the specific needs of women who have experienced sexual violence, particularly in the acute phase. This study aims to address this gap by adapting the ASSYST protocol-originally developed for trauma-related acute stress-and evaluating its utility in real-world clinical settings.

The ASSYST-VS protocol consists of five 90-minute sessions. The first session focuses on psychoeducation and emotional regulation using trauma-sensitive yoga techniques (YST) to promote safety and establish a therapeutic alliance. Sessions two through five focus on desensitizing the traumatic event using an EMDR-informed version of the ASSYST protocol adapted for this population.

Given the high risk of psychopathology following sexual violence, no control group will be included for ethical reasons. Participants will be recruited from Specialized Intervention Services (SIE) in Catalonia and CAPSEM centers in Madrid. Following informed consent, participants will complete both clinician-administered and self-report assessments measuring PTSD symptoms, anxiety, depression, sleep quality, emotional well-being, and functional capacity. All study procedures will adhere to strict confidentiality protocols and comply with the General Data Protection Regulation (GDPR).

Feasibility will be assessed through adherence and dropout rates, as well as participant satisfaction. The expected sample size (n = 36) is based on previous studies with similar interventions and was calculated using G*Power to ensure adequate statistical power.

Primary outcomes include changes in PTSD symptoms (International Trauma Questionnaire, ITQ), emotional distress (Generalized Anxiety Disorder Scale, GAD-7; Patient Health Questionnaire, PHQ-9), functional impairment (Inadaptation Scale), sleep problems (Pittsburgh Sleep Quality Index, PSQI), and well-being (Warwick-Edinburgh Mental Well-being Scale, WEMWBS). Participant satisfaction will be measured with the Client Satisfaction Questionnaire (CSQ). This project seeks to provide evidence for a scalable, early-phase trauma intervention with high clinical relevance.

ELIGIBILITY:
Inclusion Criteria:

* Be a woman aged 18 or older
* Have experienced at least one episode of sexual violence within the past 6 months
* Be currently receiving care from one of the following centers:
* Servei d'Intervenció Especialitzada (SIE) in Garraf-Penedès or Baix Llobregat (Catalonia)
* CAPSEM Norte or CAPSEM Sur (Madrid)
* Present acute post-traumatic stress symptoms (score > 0 on items 3.1 to 3.5 of the Trauma Screening Questionnaire - TSQ)
* Be capable and willing to provide informed consent
* Be fluent in Spanish or Catalan The intervention is offered under the assumption that women seeking support from specialized services are in need of early psychological intervention, and may benefit from a brief trauma-focused approach. This inclusive design seeks to maximize access to care and promote recovery in real-world settings.

Exclusion Criteria:

* Active substance abuse that would interfere with treatment participation
* Intellectual or cognitive disability that prevents completion of the intervention protocol
* Active suicidal ideation at the time of the intervention
* Inability to communicate in Spanish or Catalan

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Only individuals who identify as women are eligible to participate in this study. This means that the study is specifically designed for women due to the nature of the support services involved and the specific focus on experiences of sexual violence. Participants must be 18 years of age or older and currently receiving care from the Specialized Intervention Service in Gender-Based Violence (SIE) in the Garraf/Penedès region of Barcelona, which is part of the Department of Feminisms and Equality of the Government of Catalonia.
Enrollment: 36 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in posttraumatic stress symptoms | Before the intervention (baseline) Immediately after the intervention (3 weeks) 3-month follow-up
  International Trauma Questionnaire (ITQ; Cloitre et al., 2018) Post-Traumatic Stress Disorder (PTSD) and Complex PTSD (CPTSD) symptoms based on ICD-11 criteria.
  Administration: Self-administered online via a Qualtrics link. Interpretation: Higher scores indicate greater symptom severity of PTSD and CPTSD

SECONDARY OUTCOMES:
Changes in anxiety symptoms | Baseline Post-intervention (3 weeks) 3-month follow-up
  Generalized Anxiety Disorder-7 (GAD-7; Spitzer et al., 2006; Spanish version by García-Campayo et al., 2010) Symptoms of generalized anxiety experienced over the past two weeks. Administration: Self-administered online with support available if needed. Interpretation: Higher scores indicate greater levels of generalized anxiety.
Changes in depression symptoms | Baseline Post-intervention (3 weeks) 3-month follow-up
  Patient Health Questionnaire-9 (PHQ-9; Kroenke et al., 2001; Spanish version by Díez-Quevedo et al., 2001) Depressive symptoms experienced over the past two weeks. Administration: Self-administered via Qualtrics. Interpretation: Higher scores indicate more severe depressive symptoms.
Changes in sleep dimensions | Baseline Post-intervention (3 weeks) 3-month follow-up
  Pittsburgh Sleep Quality Index - Short Version (PSQI; Buysse et al., 1989) Sleep quality and patterns, including sleep duration, latency, efficiency, disturbances, and daytime dysfunction.
  Administration: Self-administered. Interpretation: Higher scores indicate poorer sleep quality.
Changes in general Impairment | Baseline Post-intervention (3 weeks) 3-month follow-up
  General Impairment Index (Índice de Inadaptación General; Echeburúa, Corral & Fernández-Montalvo, 2000) The degree of functional impairment or maladjustment in daily life, including personal, social, and work domains.Administration: Self-administered online, with professional assistance if necessary.
  Interpretation: Higher scores reflect greater difficulties in daily functioning.
Changes in wellbeing | Baseline Post-intervention (3 weeks) 3-month follow-up
  Warwick-Edinburgh Mental Wellbeing Scale (WEMWBS; Tennant et al., 2007) Positive mental wellbeing, including positive affect, psychological functioning, and interpersonal relationships.
  Administration: Self-administered via Qualtrics. Interpretation: Higher scores indicate better mental wellbeing.
Satisfaction with the intervention | Only after the intervention (3 weeks)
  Client Satisfaction Questionnaire-8 (CSQ-8; Attkisson & Zwick, 1982) Participant satisfaction with the intervention, including perceived effectiveness, quality, and willingness to recommend.
  Administration: Self-administered online. Interpretation: Higher scores indicate greater satisfaction with the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Valiente, Full Porfessor, Principal Investigator — Universidad Complutense de Madrid; Yolanda Ballesteros Gonzalez, PhD student, Principal Investigator — Universidad Complutense de Madrid; Regina Espinosa, Full Porfessor, Principal Investigator — Camilo Jose Cela University
Locations (1):
- Universidad Complutense de Madrid, Madrid, Pozuelo de Alarcón, Spain

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol Statistical Analysis Plan (SAP) Informed Consent Form (ICF) Clinical Study Report (CSR) Analytic Code
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code